CLINICAL TRIAL: NCT05865860
Title: Application and Safety Evaluation of 3D Visualization System in Microsurgical Training
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Other Study IDs: 2022KYPJ220
Record Dates: First submitted 2023-03-28; First posted 2023-05-19 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-01

CONDITIONS: Microsurgery; Binocular Visual Function; Nervous System
MeSH Terms: conditions — Neurologic Manifestations

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ophthalmologists with microsurgical training: Participants underwent training by digital and microscope, and we observed the changes of functions before and immediately after the training

SUMMARY:
Based on the relative shortage of ophthalmic surgeons in China, the long micromanipulation cycle and the existing micromanipulation training methods have their own limitations, such as traditional operating in porcine eyes limited to synchronous guidance and evaluation, while surgical simulators are very different for the simulation of real tissues, and the price is expensive and easy to lose. Based on these, the development of a digital training system, that is, based on traditional micromanipulation platforms such as animal tissue, physical microscopic instruments supplemented by synchronous surgical guidance and evaluation, can combine the advantages of traditional training and simulator, so as to improve the efficiency of ophthalmic surgeon training, and also provide digital ideas for other disciplines based on traditionally surgical teaching.

DETAILED DESCRIPTION:
The digital vision technology are required for the daily training of microsurgeons enrolled in our study. We only observed biological indicators of surgeons before and immediately after the operation using the digital technology, according with the prospective observational study design.

ELIGIBILITY:
Inclusion Criteria:

* Age:20-45 years
* Refractive diopters: spherical: - 6.00 to + 1.00 D, cylindrical: - 1.50 to - 0 D, and binocular difference less than 1.5 D
* Monocular best-corrected visual acuity (BCVA) ≥ 20/20
* Normal stereoacuity (60 s of arc or better)

Exclusion Criteria:

* history of strabismus
* history of systemic diseases
* history of eye surgery

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: ophthalmologists
Sampling Method: Non-Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-04-13 (Estimated); Study Completion 2024-04-13 (Estimated)

PRIMARY OUTCOMES:
change of accommodative lag between pre- and post- microsurgery under digital visualization system. | 5 minutes before the microsurgery and after the microsurgery within 3minutes
  Accommodative lag was measured by Monocular estimation method (MEM) retinoscopy before and immediately after the microsurgery

SECONDARY OUTCOMES:
heart rate variability | 1 minutes before the microsurgery and after the microsurgery within 1minutes
  Heart rate variability is the physiological phenomenon of variation in the time interval between heartbeats. It is measured by the variation in the beat-to-beat interval. We measure heart rate variability by a wearable watch
surgical performance | Intraoperative (When participant performs the operation, the surgical videos is simultaneously recorded.)
  Surgical videos were used to assess the microsurgical performance by modified Objective Structured Assessment of Technical Skill (OSATS) assessment tool.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China